CLINICAL TRIAL: NCT04810403
Title: An Open Trial Pilot Study of SOMEBODY, a Social Media-based Eating Disorder Prevention Program for College Women
Brief Title: SOMEBODY, a Social Media-based Eating Disorder Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Pamela Keel, Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00001960
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Eating Disorder Symptom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOMEBODY Eating Disorder Prevention Program (Experimental): All participants will be recruited to participate in the SOcial MEdia (SOME) adaptation of activities from the BODY Project (SOMEBODY).
  Interventions: Behavioral: SOMEBODY Eating Disorder Prevention Program

INTERVENTIONS:
Behavioral: SOMEBODY Eating Disorder Prevention Program — Participants will receive daily activities to complete on their most frequently used social media platform for 14 consecutive days. Daily activities have been adapted from the Body Project - an intervention that has been demonstrated to reduce internalization of the thin ideal and reduce risk for eating disorders. Examples of activities to be piloted include unfollowing social media accounts the participant perceives as reinforcing the thin-ideal and posting a selfie without makeup or editing. Based on feedback from participants, the intervention may be altered to improve acceptability, feasibility, and preliminary evidence of potential efficacy.

SUMMARY:
The purpose of this study is to develop and evaluate the feasibility, acceptability, and preliminary evidence of potential efficacy of a social-media based intervention to reduce risk factors for eating disorders in college women.

DETAILED DESCRIPTION:
Previous research supports an association between specific aspects of social media use and increased eating pathology in correlational designs and that specific aspects of social media use cause increases in risk factors for eating disorders. The aim of the current project is to determine whether social media use can be altered to cause decreases in eating disorder risk factors. To accomplish this, college women will be recruited to participate in an open trial of a pilot program that adapts activities used within evidence-based eating disorder prevention programs to be used on social media platforms. The intervention is designed to target internalization of the thin ideal.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 to 25 years old
* score in the top 50th percentile for time spent on social media each day

Exclusion Criteria:

* male
* <18 years or >25 years old
* individuals who screen positive for a Diagnostic Statistical Manual-5 eating disorder on the Eating Disorder Diagnostic Scale

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention | 2 weeks
  Acceptability will be evaluated with 7-point Likert scale ratings, with a score ≥5 indicating that participants found the intervention acceptable
Feasibility of intervention | 2 weeks
  Feasibility will be evaluated as the percentage of consented and enrolled participants who complete ≥10 of the 14 days of the intervention, with ≥80% indicating feasibility
Change in internalization of the thin ideal | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Sociocultural Attitudes Towards Appearance Questionnaire - 4 Revised (SATAQ-4R) Internalization Subscales will be used to measure internationalization of the thin ideal before and after the intervention. An effect size of d=.50 for within subject change in score will establish preliminary evidence of potential efficacy

SECONDARY OUTCOMES:
Change in body image concerns | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Eating Disorders Examination Questionnaire Weight and Shape Concerns subscales adapted for the past 7 days will be used to measure change in body image before and after the intervention
Change in dietary restraint | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Eating Disorders Examination Questionnaire Dietary Restraint subscale adapted for the past 7 days will be used to measure change in dietary restraint before and after the intervention
Change in bulimic symptoms | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Eating Disorders Examination Questionnaire Self-Reported Bulimic Symptom Composite Score adapted for the past 7 days will be used to measure change in bulimic symptom frequency before and after the intervention
Change in disordered eating | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Eating Disorders Examination Questionnaire Global Score adapted for the past 7 days will be used to measure change in disordered eating before and after the intervention
Change in social media use | Pre-intervention assessment to post-intervention assessment (or approximately 14 days from baseline)
  The Social Media Use Questionnaire items assessing frequency and type of engagement with social media will be used to measure change in social media use before and after the intervention
Adherence to protocol - self-reported | 2 weeks
  The Social Media Use Questionnaire items assessing adherence to daily social media activities will be used to measure self-reported adherence after the intervention
Adherence to protocol - observed | Daily for the 14 days of the intervention
  With participant consent, a research assistant will follow the social media account the participant plans to use for the SOMEBODY intervention and will complete a checklist on a daily basis (yes/no) on whether or not the participant completed the daily assignment

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Keel, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State University Psychology Department, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No